## The GlaxoSmithKline group of companies

**Division:** Worldwide Development **Retention Category:**GRS019

Information Type: Clinical Pharmacology Reporting and Analysis Plan

| Title: | Clinical Pharmacology Reporting and Analysis Plan for a repeat- |
|--------|-----------------------------------------------------------------|
| | dose, open-label, parallel-group study to assess the |
| | pharmacokinetics of GSK1278863 and metabolites in subjects |
| | with End Stage Renal Disease undergoing peritoneal dialysis. |

Compound Number: GSK1278863

Effective Date: 14-SEP-2017

# **Description**:

The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the Clinical Pharmacology Study Report for Protocol 200942. This study is intended to characterize the pharmacokinetics of GSK1278863 and its metabolites in subjects with end stage renal disease (ESRD) undergoing peritoneal dialysis. This document will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

**Subject:** GSK1278863, Prolyl hydroxylase inhibitor, Anemia, Chronic kidney disease, peritoneal dialysis, erythropoiesis stimulating agents, analysed in, pharmacokinetics

#### **Author's Name and Functional Area:**

| PPD | Quantitative Science India | Quantitative Science India |
|-----|----------------------------|----------------------------|
| PPD | | Quantitative Science India |
| PPD | | Quantitative Science India |

## **Approved by Email:**

The Discovery Biometrics Director (or designee) will give final approval

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF AI | BBREVIATIONS | 4 |
| 1. | INTRO | DDUCTION | 6 |
| 2. | STUD`<br>2.1. | Y OBJECTIVE(S) AND ENDPOINT(S) Study Objective(s) 2.1.1. Primary Objective(s) | <mark>7</mark> |
| 3. | STUD | Y DESIGN | 8 |
| 4. | PLANN<br>4.1.<br>4.2. | NED ANALYSESInterim AnalysesFinal Analyses | 8 |
| 5. | ANALY | YSIS POPULATIONS | 8 |
| 6. | HYPO | THESES AND TREATMENT COMPARISONS | 9 |
| 7. | GENE 7.1. 7.2. 7.3. 7.4. 7.5. | RAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING Reporting Conventions Data Management Premature Withdrawal and Missing Data Baseline Definition Derived and Transformed Data 7.5.1. Demographic and Population parameters 7.5.1.1. Study Day 7.5.1.2. Date of Birth 7.5.1.3. Age 7.5.1.4. Body Mass Index (BMI) 7.5.1.5. Exposure 7.5.2. Safety Parameters 7.5.2.1 Adverse Events 7.5.3. Change from Baseline 7.5.4. Pharmacokinetic Parameters 7.5.5. Multiple Measurements at One Timepoint Values of Potential Clinical Importance 7.6.1. Laboratory Values 7.6.2. Vital Signs. 7.6.3. ECG. | 9121212121313131314141414 |
| 8. | STUD'<br>8.1.<br>8.2.<br>8.3. | Y POPULATION Subject Disposition and Demographics Protocol Deviations Concomitant Medications | 17<br>17 |
| 9. | SAFE1<br>9.1.<br>9.2.<br>9.3. | TY ANALYSES Extent of Exposure Adverse Events Deaths and Serious Adverse Events | 18<br>19 |

| | 9.4. | Adverse Events Leading to Discontinuation of Investigational Product and/or Withdrawal from the Study and Other Significant | |
|---|---|---|---|
| | | Adverse Events | 19 |
| | 9.5. | Clinical Laboratory Evaluations | 19 |
| | 9.6. | Vital Signs and Body Weight | 19 |
| | 9.7. | Electrocardiograms | 19 |
| 10. | PHAR | MACOKINETIC ANALYSES | 20 |
| | 10.1. | | |
| | 10.2. | | 20 |
| | 10.3. | | |
| | | • | |
| 11. | PHAR | MACODYNAMIC/BIOMARKER ANALYSES | 24 |
| 12 | PΗΔR | MACOGENETIC ANALYSIS | 24 |
| 12. | 1 11/413 | WIAGOGENETIC ANALTOIC | 27 |
| 13. | REFE | RENCES | 25 |
| 14. | ATTA | CHMENTS | 26 |
| | 14.1. | Table of Contents for Data Display Specifications | 26 |
| | | 14.1.1. Study Population | 27 |
| | | 14.1.2. Safety Tables | 28 |
| | | 14.1.3. Pharmacokinetic Figures and Tables | 30 |
| | | 14.1.4. Pharmacodynamic Figures and Tables | |
| | | 14.1.5. ICH Listings | |
| | | 14.1.6. Other Listings | 39 |
| | 14.2. | Data Display Specifications (Example Shells) | 40 |

# **LIST OF ABBREVIATIONS**

| AE | Adverse Event |
|---|---|
| ALT | Alanine aminotransferase (SGPT) |
| ANOVA | Analysis of Variance |
| APD | Ambulatory Peritoneal Dialysis |
| AST | Aspartate aminotransferase (SGOT) |
| AUC | Area under concentration-time curve |
| | Area under the concentration-time curve from time zero (pre-dose) |
| $AUC (0-\infty)$ | extrapolated to infinite time |
| %AUCex | Percentage of AUC (0-\infty) obtained by extrapolation |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to |
| | last time of quantifiable concentration |
| AUC (0-τ) | Area under the concentration-time curve over the dosing interval |
| BMI | Body mass index |
| BP | Blood pressure |
| BPM | Beat Per Minute |
| BQL | Below the quantification limit |
| BUN | Blood urea nitrogen |
| CAPD | Continuous Ambulatory Peritoneal Dialysis |
| CBC | Complete blood count |
| Cmax | Maximum observed concentration |
| IDMC | |
| IDSL | Independent Data Monitoring Committee Integrated Data Standards Library |
| IU | Integrated Data Standards Library International Unit |
| IV | Intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | |
| mL | Milligrams Milliliter |
| MRT | Mean residence time |
| MSDS | Material Safety Data Sheet |
| | Milliseconds |
| msec<br>NQ | Non-quantifiable concentration measured as below LLQ |
| PD | Pharmacodynamic |
| PGx | , |
| PK | Pharmacogenetics Pharmacokinetic |
| PSRI | Periodic Safety Reports for Investigators |
| QC | Quality control |
| QD | Once daily |
| RAP | Reporting and Analysis Plan |
| t OR tlast | Time of last observed quantifiable concentration |
| t <sup>1</sup> / <sub>2</sub> | Terminal phase half-life |
| τ | Dosing interval |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| tmax | Time of occurrence of Cmax |

200942

| ULN | Upper limit of normal |
|-----|-----------------------|
| WBC | White blood cells |

# **Trademark Information**

| Trademarks of the GlaxoSmithKline group of companies |
|------------------------------------------------------|
| HARP |

| Trademarks not owned by the GlaxoSmithKline group of companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Pharmacology Study Report for Protocol 200942:

| Revision Chronology: Protocol | | |
|-------------------------------|-------------|-----------------|
| 2013N179529_00 | 2014-APR-11 | Original |
| 2013N179529_01 | 2014-JUN-06 | Amendment No. 1 |
| 2013N179529_02 | 2014-JUN-24 | Amendment No. 2 |
| 2013N179529_03 | 2014-JUL-01 | Amendment No. 3 |
| 2013N179529_04 | 2014-DEC-12 | Amendment No. 4 |
| 2013N179529_05 | 2015-SEP-10 | Amendment No. 5 |
| 2013N179529_06 | 2016-JUN-20 | Amendment No. 6 |

All decisions regarding final analysis, as defined in this RAP document, have been made prior to Database Freeze (unblinding) of the study data.

# 2. STUDY OBJECTIVE(S) AND ENDPOINT(S)

# 2.1. Study Objective(s)

# 2.1.1. Primary Objective(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| Characterize the steady-state PK of GSK1278863 and metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), GSK2531401 (M13) in ESRD subjects undergoing peritoneal dialysis | • [AUC(0-τ), AUC (0-∞)] (Day 1 only), and Cmax of GSK1278863 and metabolites on Day 1 and Day 14 |
| Secondary | |
| Evaluate the safety and tolerability of GSK1278863 in ESRD subjects undergoing peritoneal dialysis | • Subject incidence of treatment emergent adverse events, including clinically-significant changes in physical exams, laboratory safety tests, ECG and vital signs |
| Characterize the peritoneal dialysis clearance of GSK1278863 and metabolites in ESRD subjects undergoing peritoneal dialysis | <ul> <li>Peritoneal dialysis clearance, tmax and t½ of GSK1278863 and metabolites on Day 1 and Day 14</li> <li>Accumulation ratio and time invariance ratio (as data permit) of GSK1278863 and metabolites</li> </ul> |
| Characterize the plasma profile of erythropoietin and hepcidin after repeat dose administration of GSK1278863 in ESRD subjects undergoing peritoneal dialysis | Erythropoietin and hepcidin plasma<br>concentrations |
| Exploratory | |
| Characterize the plasma protein binding of steady-state GSK1278863 and select metabolites in ESRD subjects undergoing peritoneal dialysis | Steady-state GSK1278863 and<br>metabolite unbound concentration and<br>free fraction |
| Characterize the effect of different peritoneal dialysis solutions on GSK1278863 and metabolites in ESRD subjects undergoing peritoneal dialysis | Descriptive summary of GSK1278863<br>and metabolite PK by different<br>peritoneal dialysis solutions utilized |

# STUDY DESIGN

This is a repeat-dose, open label, 2 cohort study to assess the pharmacokinetics of GSK1278863 and metabolites in ESRD subjects undergoing peritoneal dialysis. GSK1278863 (5 mg) will be orally administered once daily for 14 days to approximately 12 ESRD subjects;

- Cohort 1 will enrol subjects on continuous ambulatory peritoneal dialysis (CAPD) to complete all dosing and critical assessments
- Cohort 2 will enrol subjects on automated peritoneal dialysis (APD) to complete all dosing and critical assessments.

Further details about the study design can be found in Section 3 of the protocol.

## 4. PLANNED ANALYSES

# 4.1. Interim Analyses

 Informal PK reviews will be conducted throughout the study to assist Phase III development of the compound

# 4.2. Final Analyses

The final planned analyses will be performed after all subjects have completed the study and after database freeze. See Section 8 to Section 10 for all final planned analyses for this study.

# 5. ANALYSIS POPULATIONS

## **All Screened Population**

The "All Screened" population will be defined as all subjects screened.

## **Enrolled Population**

All participants who were enrolled for the trial and for whom a record exists on the study database.

## **All Subjects Population**

Any subject enrolled into the study who receives at least one dose of study medication will be included in the 'All Subjects' Population. This will be the population used for the study population and safety analyses.

## **Pharmacokinetic Population**

The 'PK Population' is defined as subjects in the 'All Subjects' population for whom a pharmacokinetic sample was obtained and analysed. This will be the population used for the Pharmacokinetic displays.

# 6. HYPOTHESES AND TREATMENT COMPARISONS

## **Precision Estimation**

This study is designed to estimate pharmacokinetic endpoints of GSK1278863 and metabolites in ESRD patients undergoing peritoneal dialysis following repeat administration of 5 mg once daily GSK1278863.

There will be two cohorts of subjects in this study: subjects with CAPD and subjects with APD.

No formal statistical hypotheses will be tested. An estimation approach will be used to evaluate the comparisons of interest, with point estimates and associated 90% confidence intervals presented to provide a range of plausible values for the comparisons.

Table 1 Treatment and Other Sub-Group Descriptions for Data Displays

| Randomisation | | Final Data Display<br>(i.e. HARP / other) |
|---|---|---|
| Treatment | Cohort Description | Cohort |
| 5 mg GSK1278863 | Continuous Ambulatory<br>Peritoneal Dialysis | CAPD |
| | Automated Peritoneal Dialysis | APD |

# 7. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING

# 7.1. Reporting Conventions

- All data displays will be presented according to the Integrated Data Standards Library (IDSL) reporting standards, where applicable. In general, data will be listed by cohort, subject, and time point and summarized by cohort (i.e. by CAPD, APD and combined) and time point
- Analyses will be performed using the 9.1.3 version of the SAS System or higher (SAS is a registered trademark of the SAS Institute Inc., Cary, NC, USA).
   Programs will be imported into HARP and the final output will be produced by running drivers in HARP.
- Data collected at unplanned (i.e. unscheduled) time points will not be included in the summaries by visit unless otherwise stated. Unscheduled or unplanned readings will be presented in the listings and they will be included when determining worst-case flagging for post-baseline summaries.

- In all data displays, planned and actual relative times will be relative to the study drug dosing time of the relevant dosing session.
- Planned times relative to study drug dosing will be used in all summary tables and summary (mean and median) figures.
- Actual times relative to study drug will be used in all listings and individual PK figures.
- Refer to IDSL standards (when applicable) for decimal place conventions. Raw data will generally be presented to the same number of decimal places as it was collected.
- All data will be reported according to the actual treatment the subject received.
   Any departures from the planned treatment according to the randomization schedule will be documented in the report.
- All observations that occurred prior to dosing will be considered as part of the pre-dose period. All observations that occur during dosing will be attributed to the subject's treatment. Observations occurring after 28 days after the last dose of study medication will not be recorded in the database.
- Deviations from the analyses in the RAP will be identified in the final clinical pharmacology study report.

# 7.2. Data Management

| Data Type | Source | Format of Data | Planned Date of Final File <sup>1</sup> | Responsibility |
|---|---|---|---|---|
| Safety | SDTM datasets | CDISC | DBF | CPDS |
| Biomarker | External CRO | CSV file | DBF+X <sup>4</sup> days | CPDS |
| SDTM PC | PK concentration data merged with SI PK | CDISC | DBF + X Days | SDTM Conversion<br>Service (SCS) |
| Winnonlin file<br>created from<br>ADPC (PK<br>Conc) | Analysis Dataset for PK Concentrations | CSV file | SDTM PC + X <sup>4</sup> Days | QSI (Prog) |
| PK Parameter | Winnonlin-<br>posted to HARP<br>by CPMS <sup>3</sup> | CSV file | PK Conc Winnonlin<br>+ X <sup>4</sup> days <sup>2</sup> | CPMS |
| SDTM PP | PK parameter data | CDISC | PK Parameter<br>Winnonlin + X <sup>4</sup><br>days <sup>2</sup> | SDTM Conversion<br>Service (SCS) |

<sup>1.</sup> This is for study teams to determine upfront if there is a possibility of not meeting the completion of the CPSR within 6 months of LSLV (i.e. novel data that may not be available until several months after LSLV).

<sup>2.</sup> Provided source data is clean.

<sup>3.</sup> PK concentration data is released via SMS2000 by DMPK and the SI PK dataset contains date/times and PK sample ID.

<sup>4.</sup> Standard timelines are not followed for this study.

# 7.3. Premature Withdrawal and Missing Data

All subjects who withdraw prematurely from the study/study drug will be documented and the reason for their withdrawal recorded in the final Clinical Pharmacology Study Report (CPSR). All available data from subjects who withdraw will be listed and all available planned data will be included in the summaries according to the populations defined in Section 5.

In the event that the study is prematurely discontinued, all available data will be listed and a review carried out by the study team to assess which statistical analyses are still considered appropriate.

# 7.4. Baseline Definition

The following table indicates the baseline day to be used in any change from baseline listings / summaries / graphical presentations or as a covariate in a statistical analysis:

| Parameter | Baseline Days Collected | | | Baseline To Be |
|---|---|---|---|---|
| | Screening | <b>Day -1</b> | Day 1 Predose | Used in Analysis |
| | | | | / Summaries |
| Safety: | | | | |
| ECG | X | X | | Day -1 |
| Vital Signs | X | X | | Day -1 |
| Lab | X | X | | Day -1 |
| EPO, Hepcidin | | | X | Day 1 Predose |

# 7.5. Derived and Transformed Data

## 7.5.1. Demographic and Population parameters

## 7.5.1.1. Study Day

Study day will be calculated as number of days from baseline date, as outlined below:

```
ScenarioStudy Dayreference date is missingstudy day = missingreference date < IP start date</td>study day = reference date − IP start datereference date ≥ IP start datestudy day = reference date − (IP start date + 1)
```

#### 7.5.1.2. Date of Birth

Note that only the year of birth has been captured, so all dates of birth are 30<sup>th</sup> June XXXX, where XXXX is the year of birth.

## 7.5.1.3. Age

Age is calculated based on screening date, using date of birth, truncated to integer value. Note that only the year of birth has been collected where the day and month would be 30<sup>th</sup> June for all patients. Therefore, the derivation of age will be approximate.

The derivation of age will be footnoted on appropriate displays.

## 7.5.1.4. Body Mass Index (BMI)

Body Mass Index (BMI) is calculated as follows:

BMI = weight in kg /  $(\text{height in cm})^2$ 

#### 7.5.1.5. Exposure

Exposure is calculated as follows:

Study Drug Exposure (days) = (Treatment Stop Date – Treatment Start Date) + 1

# 7.5.2. Safety Parameters

## 7.5.2.1. Adverse Events

Note that the database has been designed such that AE Onset date is missing, unknown or complete; a partial/incomplete AE onset date will be considered as missing.

#### ΑE

| AE Onset Time since First Dose | = AE Onset Date – Treatment Start Date (if treatment |
|---|---|
| | start date > AE onset date) |
| | = AE Onset Date – Treatment Start Date + 1 (if |
| | treatment start date <= AE onset date) |
| | = missing otherwise |
| AE Duration (in days) | = AE Resolution Date – AE Onset Date + 1 |
| AE is "On Treatment" | if the AE onset date is on or after the treatment start |
| | date and on or before the treatment stop date |
| AE is "Post-Treatment" | if the AE onset date is after the treatment stop date |
| AE is considered drug-related | if the relationship is marked 'Yes' on the case report |
| _ | form, or the value is missing |

# 7.5.3. Change from Baseline

The change from baseline will be calculated by subtracting the baseline values from the individual post-randomisation values. If either the baseline or post-randomisation value is missing, the change from baseline is set to missing as well.

#### 7.5.4. Pharmacokinetic Parameters

For the purposes of calculating summary statistics and for statistical analysis, all PK parameters with the exception of tmax will be loge transformed.

Between subject coefficient of variation CV<sub>b</sub> (%) will be calculated according to the following methods:

Untransformed Data : 100 \* (SD/Mean) where SD is the standard deviation of the untransformed data

Transformed Data  $: SQRT(exp(SD^2-1)) * 100$ where SD is the standard deviation of the  $log_e$ -transformed data.

# 7.5.5. Multiple Measurements at One Timepoint

Where multiple measurements are recorded for a particular time point, the mean of the measurements will be calculated and used in any derivation of summary statistics. However, all available data will be listed.

Where more than the specified number of measurements has been taken, the most recently recorded values will be used in the derivation of the appropriate summary measure (i.e. mean or maximum).

# 7.6. Values of Potential Clinical Importance

The following tables display the ranges to be used for flagging values of potential clinical importance for various parameters. These values will be flagged on the listings.

# **Laboratory Values of Potential Clinical Importance (Renal Failure)**

## 7.6.1. Laboratory Values

| Laboratory Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Low Flag | High Flag |
| Albumin | g/L | < 30 g/L | >55 g/L |
| Aspartate Aminotransferase | IU/L | | ≥3x ULRR |
| Alanine Aminotransferase | IU/L | | ≥3x ULRR |
| Bilirubin (total and direct/indirect) | μmol/L | | ≥2x ULRR |
| Calcium | mmol/L | > 0.5 mmol/L<br>below LLRR | > 0.25 mmol/L above<br>ULRR |
| Glucose, fasting | mmol/L | <3.9 | >22 |
| Sodium | mmol/L | <130 | >150 |

| Laboratory Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Low Flag | High Flag |
| Total CO2 | mmol/L | <20 | >32 |
| GGT | IU/L | | >=2ULRR |
| Alkaline phosphatase | IU/L | | >=3xULRR |
| Uric Acid | Mg/dL | | >6.0 mg/dL |
| Total Protein | IU/L | <llrr< td=""><td>&gt;15 g/L bove ULRR</td></llrr<> | >15 g/L bove ULRR |
| Potassium (serum) | mmol/L | > 0.5 mmol/L<br>below LLRR | > 1.0 mmol/L above<br>ULRR |

| Laboratory Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Low Flag (< x) | High Flag (>x) |
| Hemoglobin | g/dL | < 7.5 | >=13.0 |
| Platelet Count | GI/L | < 80x GI/L | > 500x GI/L |
| WBC Count | GI/L | > 1x GI/L below<br>LLRR | >5x GI/L above<br>ULRR |
| Neutrophils | GI/L | < 0.5x LLRR | |
| Lymphocytes | GI/L | < 0.5x LLRR | |

| Laboratory Parameter | Units | Clinical Concern Range | |
|----------------------|-------|------------------------|----------------|
| | | Low Flag (< x) | High Flag (>x) |
| Ferritin | ng/mL | | > 1200 |
| TSAT | % | <15 | >40 |

## 7.6.2. Vital Signs

| Vital Sign Parameter Units | | Clinical Concern Range | |
|----------------------------|------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≤85 | ≥180 |
| Diastolic Blood Pressure | mmHg | ≤45 | ≥110 |
| Heart Rate | bpm | ≤40 | ≥110 |

#### Notes:

- At visits where BP and HR are assessed in triplicate, the average of the 3 values will be used to assess PCI criteria.
- For subjects who undergo in-clinic dialysis, the post-dialysis BP and HR values will be used to assess PCI criteria, unless otherwise specified.

#### 7.6.3. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute QTc interval | msec | | >480 if with bundle branch block |
| Change from Baseline | | | |
| QTcB or QTcF | msec | | >60 msec |

# 8. STUDY POPULATION

It was initially expected that 30 subjects (15 in each cohort) would be needed to be recruited in order to ensure that at least 12 subjects (6 in each cohort) completed the trial. However, during the informal review of the available PK data it was determined that there were no clinically-significant differences in PK between the CAPD/APD and CKD populations, therefore the planned number of subjects was reduced to enrol 7 subjects and 5 subjects completed the study in order to minimize unnecessary additional subject exposure.

Study population data will be summarised by, or under the direct auspices of, Clinical Statistics, GlaxoSmithKline.

The precise format and content of Study Population tables and listings are shown in Section 14.1.1 and Section 14.1.5 of the RAP.

The tables will use the "All Subjects" population unless otherwise specified.

# 8.1. Subject Disposition and Demographics

A listing of subject withdrawals will include all subjects who prematurely discontinued from the study. This listing will include the discontinuation information for each subject, if there are any, including dates of discontinuation and reason for premature discontinuation. The number of subjects who completed, withdrew, and reasons for withdrawal will be tabulated.

A listing indicating whether a subject was included in each of the analysis populations will be prepared. The number of subjects included in each analysis population will be tabulated.

Demographic and racial data will be summarized using the "All Subjects" population.

## 8.2. Protocol Deviations

As outlined in the protocol deviation plan the protocol deviations will be discussed and reviewed by the study team. The frequency of the review may be amended dependent on the outcome of the initial reviews. Any protocol deviations identified will be entered into InForm eCRF. Prior to each review the DQL will run the protocol deviation check log and protocol deviation log report in InForm, discrepancies will be resolved and the report issued to the reviewing study team.

All protocol deviations that are data based will be listed.

#### 8.3. Concomitant Medications

All medications will be coded using the GSK Drug dictionary. Medications will be classified into preferred term and body system, using the GSK-Drug Anatomical Therapeutic Clinical (ATC) classification. ATC level 1 (the body system) will be shown. Medications will be sorted in descending order of total incidence across treatment groups for the ATC level 1 and in descending order of total incidence for the preferred term within each ATC level.

Medications will be defined as follows, where it should be noted that a medication can be counted in more than one phase:

| Prior | - any medication taken up to, but not including, the start date of study medication (pre-treatment phase). Therefore, prior medications have stopped prior to the subject taking study medication. |
|---|---|
| Concomitant | <ul> <li>if a medication is started or stopped on the same day of taking the first or last dose of randomised investigational product then this will be considered a concomitant medication (on-treatment phase)</li> <li>any medication started before last day in the study and the drug stop date is either missing or on or after treatment start date</li> <li>any medication with start date missing yet the stop date is on or after treatment start date</li> <li>if both start and stop dates are missing the drug is specifically indicated as continuing in the trial.</li> </ul> |
| Post study | - any drug with start date on or after last day in the study will be considered post-study drug. This will not be summarized with concomitant drugs but will be included in data listing. |

In situations where the concomitant medication status of the drug cannot be determined, available relevant information will be reviewed on a case-by-case basis to determine the status whether it should be considered 'concomitant' or 'post-study' by Clinical; the decision of the clinical group will be considered final. However, if such determination cannot be made unambiguously, the medication will be considered concomitant.

Concurrent medications will be listed, and summarized by generic term, if more than 20 concomitant medications were used.

## 9. SAFETY ANALYSES

Safety data will be summarised and listed by, or under the direct auspices of Clinical Statistics, GlaxoSmithKline.

The precise format and content of Safety tables, ICH and Other listings are shown in Section 14.1.2, Section 14.1.5 and Section 14.1.6 of the RAP.

The tables will use the "All Subjects" population unless otherwise specified.

# 9.1. Extent of Exposure

A listing of exposure data will be a by-subject listing including the cohort, treatment administered with the dates and times of treatment administration.

#### 9.2. Adverse Events

All adverse events (AEs) will be coded and classified according to system organ class, high level term, and preferred term using GSK MedDRA. All AEs will be listed. A listing of subject numbers for individual AEs will also be prepared. A summary, overall and by treatment, of the number and percent of subjects reporting each event at least once will be generated for all AEs and also for drug-related AEs. A listing of the relationship of AE body systems, group terms and verbatim text will also be produced.

#### 9.3. Deaths and Serious Adverse Events

In addition to the listing described above, deaths and serious AEs (SAEs), if they occur, will also be listed and summarized separately.

# 9.4. Adverse Events Leading to Discontinuation of Investigational Product and/or Withdrawal from the Study and Other Significant Adverse Events

If any subject withdraws due to an AE, then a listing and a summary by treatment will be provided for these subject(s).

# 9.5. Clinical Laboratory Evaluations

A listing for hematology and clinical chemistry values of potential clinical importance as described in Section 7.6, will be produced where applicable.

For hematology and clinical chemistry data, descriptive summaries for actual values by time point will be produced. A summary of urinalysis dipstick data and a listing of urinalysis data will be produced.

# 9.6. Vital Signs and Body Weight

Listing of vital signs values of potential clinical importance as described in Section 7.6, will be produced where applicable. Descriptive summaries for absolute and change from baseline values for vital signs by time point will be produced.

# 9.7. Electrocardiograms

Descriptive summaries for absolute and change from baseline values of ECG values by time point will be produced.

ECG findings will be summarized with the highest (worst) severity across replicated assessments at the specified time point used.

ECG abnormalities of clinical significance, if they occur, will be listed for each subject.

## 10. PHARMACOKINETIC ANALYSES

The reconciliation of the PK Case Report Form (CRF) and SMS2000 data will be performed by, or under the direct auspices of, Clinical Pharmacology Data Sciences (CPDS), GlaxoSmithKline.

The merge of PK concentration data, randomisation and CRF data will be performed by, or under the direct auspices of, QSI (Programmer), GlaxoSmithKline.

Derivation of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline.

Statistical analysis of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Statistics, GlaxoSmithKline.

The precise format and content of PK tables, figures, and listings are shown in Section 14.1.3 and Section 14.1.6 of the RAP.

# 10.1. Drug Concentration Measures

Concentrations of GSK1278863 and its metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), GSK2531401 (M13)) in plasma will be listed and summarized by cohort (i.e., CAPD, APD and both combined) and nominal time. Standard summary statistics will be calculated (i.e. mean, standard deviation, median, minimum and maximum). Refer to the PK Guidance document, GUI\_51487 (3.0), for more information regarding the treatment of plasma concentrations below the assay's lower limit of quantification (NQ). Individual plasma concentration-time profiles and median/mean profiles by treatment cohort will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot). See Section 14.1.3 and Section 14.1.5 Pharmacokinetic Source Figures and Tables for details.

GSK1278863 and metabolite protein binding (as a percentage) will be presented in tabular form and will be summarized descriptively. Metabolite-to-parent exposure ratios (corrected for molecular weight) will also be calculated and summarized descriptively.

Volume of drained dialysate plus concentrations and amounts of GSK1278863 and its metabolites (GSK2391220(M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), GSK2531401 (M13)) in the dialysate will be listed and summarized by cohort (i.e., CAPD, APD and both combined).

# 10.2. Deriving and Summarizing Pharmacokinetic Parameters

From the plasma concentration-time data of parent GSK1278863 and metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6) and GSK2531401 (M13)), the following pharmacokinetic parameters will be determined, as data permit:

**Day 1**: Maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve  $AUC(0-\tau)$  and  $AUC(0-\infty)$ , and apparent terminal phase half-life (t½).

**Day 14**: Cmax, tmax, AUC(0- $\tau$ ), and apparent terminal phase half-life (t½). AUC(0- $\infty$ ), AUC(0- $\tau$ ), and Cmax following single (Day 1) and repeat doses (Day 14) will be used for determination of accumulation and time-invariance ratios.

**Day 12 to 15**: Trough concentration (Ctau, or  $C\tau$ ) samples collected on Days 12 to 15 will be used to assess attainment of steady state.

- Note, to comply with CDISC reporting requirements, the following parameters also will be determined:
  - o Tlast
  - Where t½ and/or AUC(0-∞) have been derived the following parameters should also be included in the PKPAR file: No\_points\_lambda\_z, Lambda\_z\_lower, Lambda\_z\_upper, Tlast
  - If partial areas have been calculated, the following parameters should also be reported (if not included as above): No\_points\_lambda\_z, Lambda\_z\_lower, Lambda\_z\_upper

Other Plasma PK Analyses: GSK1278863 and select metabolite (GSK2487818 (M4), GSK2506102 (M5)) unbound concentration and free fraction (as a percentage) will be presented in tabular form and will be summarized descriptively. Metabolite-to-parent exposure ratios (corrected for molecular weight) will also be calculated and summarized descriptively.

• Percent protein bound will be calculated using the formula:

% Bound = (Concentration in plasma – Concentration in ultrafitrate) \* 100 / Concentration in plasma

• **Metabolite to parent ratios:** (GSK2391220(M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6) and GSK2531401 (M13)) (metabolites, M) to GSK1278863 (parent) AUC and Cmax ratios will be determined (as a percentage, including a correction for molecular weight, Mr), for example:

M: GSK1278863 % = 100\* (AUC<sub>M</sub>/AUC<sub>GSK1278863</sub>) \* (Mr<sub>GSK1278863</sub>/Mr<sub>M</sub>)

Parameters to be used in this calculation are:

Day 1: Cmax, AUC(0- $\tau$ ), AUC(0- $\infty$ )

Day 14: Cmax,  $AUC(0-\tau)$ 

Molecular weights for compounds are:

| Compound | Molecular Weight (g/mol) |
|------------------|--------------------------|
| GSK1278863 | 393.442 |
| GSK2391220 (M2) | 425.442 |
| GSK2506104 (M3) | 425.442 |
| GSK2487818 (M4) | 425.442 |
| GSK2506102 (M5) | 425.442 |
| GSK2531398 (M6) | 425.442 |
| GSK2531401 (M13) | 441.442 |

• **Percent drug related marterial (%DRM):** will be determined for parent as well as each metabolite, where the denominator is the sum of the exposures of all analytes. Where all these AUCs are corrected for molecular weight (Mr).

## Example:

$$\%DRM_{GSK1278863} = 100*AUC_{GSK1278863} / (AUC_{GSK1278863} + AUC_{M2} + AUC_{M3} + AUC_{M4} + AUC_{M5} + AUC_{M6} + AUC_{M13}).$$

Parameters to be used in this calculation are:

Day 1: AUC(0- $\tau$ ), AUC(0- $\infty$ )

Day 14:  $AUC(0-\tau)$ 

 Peritoneal dialysis clearance of GSK1278863 and metabolites will be calculated from Day 14 dialysate excretion data as total amount of analyte excreted over 24 h divided by plasma AUC(0-τ).

$$CLd = Ae(0-\tau) / AUC(0-\tau)$$

where Ae is the amount of analyte excreted in dialysate over the 24 h dialysate collection period

Ae = total dialysate volume \* dialysate concentration

All the derived parameters described above will be listed. For each of these parameters, except t<sub>max</sub>, the following summary statistics will be calculated for each cohort (CAPD,APD and combined) as well as different peritoneal dialysis solution (number of categories to be determined): median, maximum, minimum, arithmetic mean, standard deviation, coefficient of variation, geometric mean, 95% confidence interval for the

geometric mean and standard deviation of logarithmically transformed data. For  $t_{max}$ , median, maximum, minimum, arithmetic mean and standard deviation will be calculated. The first point, last point and number of points used in the determination of  $\lambda_z$  will be included on the listing of the derived parameters.

# 10.3. Statistical Analyses

Descriptive statistics (n, arithmetic mean and associated 95% confidence interval, standard deviation, minimum, median, maximum) will be calculated for all pharmacokinetic endpoints of GSK1278863 and metabolites by Cohort. In addition geometric means, associated 90% CIs, and estimates of between-subject CVs (CVb (%)), will be calculated for each Cohort where

Geometric mean=exp (mean on log<sub>e</sub> scale)

CVb (%)=SQRT(exp(SD\*\*2)-1)x100, where SD is the standard deviation of the loge-transformed data.

## **Steady State Assessment**

Trough concentration ( $C\tau$ ) samples collected on the specified days (Days 12, 13, 14, and the 24 h post-dose sample on Day 14) will be used to assess attainment of steady state. Individual trough concentration data  $C\tau$  will be plotted and listed.  $C\tau$  will be summarized by day and cohort, and the mean and median plots will be provided.

Steady state will be assessed separately for GSK1278863 and metabolites in each cohort.

A linear mixed effects ANOVA model will be used to evaluate steady state for GSK1278863 and each metabolite. The dependent variable will be log-transformed Predose (trough) concentrations ( $C\tau$ ) on Days 12 to 15. Independent variables in the model include day (as a continuous variable) as a fixed effect and subject as a random effect.

Assessment of plasma GSK1278863 and metabolites steady state will be assessed by evaluating the estimated slope for the day parameter and associated 90% CI for both the cohorts combined.. A steady state attainment is defined as the 90% confidence interval of the slope including 0.

## **Secondary Comparisons:**

#### **Assessment of Accumulation**

To estimate the extent of accumulation for GSK1278863 and metabolites after repeat dosing, the observed accumulation ratio R0 will be determined.

$$R_0 = \frac{AUC(0-\tau)_{ss}}{AUC(0-\tau)}$$

Where AUC(0- $\tau$ )ss is AUC from time zero to t h under steady state and AUC (0 - $\tau$ ) is AUC from time zero to dosing interval at Day 1.

To evaluate the accumulation ratio, statistical analysis of GSK1278863 and metabolite PK data for each cohort will be performed separately after a log transformation of the data.

A mixed effect model will be fitted with day (single and repeat dose), as fixed effects and subject as a random effect. Day 14 will be compared to Day 1 in order to estimate the accumulation ratios, Ro= (AUC (0- $\tau$ , Day14): AUC (0- $\tau$ , Day1). The ratios will be calculated by back-transforming the difference between the LS means.

Using the pooled estimate of variance, 90% confidence intervals will be calculated for the primary comparisons, and back-transformed to the original scale.

## **Assessment of Time Invariance**

To evaluate the time invariance ratio, statistical analysis of (AUC  $(0-\infty)$  Day 1) and AUC  $(0-\tau)$  (Day14), of GSK1278863 and metabolites for each cohort will be performed separately after a log transformation of the data.

A mixed effect model will be fitted with day as a fixed effect and subject as a random effect. Day 14 AUC  $(0-\tau)$  will be compared to Day 1 AUC  $(0-\infty)$  in order to estimate the time invariance ratios, RS= AUC  $(0-\tau)$ , Day 14: AUC  $(0-\infty)$ , Day 1). The ratios will be calculated by back-transforming the difference between the LS means.

Using the pooled estimate of variance, 90% confidence intervals will be calculated for the primary comparisons, and back-transformed to the original scale.

## 11. PHARMACODYNAMIC/BIOMARKER ANALYSES

Plasma erythropoietin and hepcidin concentrations will be presented in graphical and/or tabular form and will be summarized descriptively. The concentration values will be listed by cohort, subject, and time point and will be summarized by cohort and time point.

## 12. PHARMACOGENETIC ANALYSIS

Samples will be collected and stored. No prospective analyses will be performed.

# 13. REFERENCES

GlaxoSmithKline Document Number 2013N179529\_03 Study ID 200942. A repeat-dose, open-label, parallel-group study to assess the pharmacokinetics of GSK1278863 and metabolites in subjects with End Stage Renal Disease undergoing peritoneal dialysis. (Effective date: 01-JUL-2014)

Schuirmann DJ. 1987. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability, J Pharmacokinetic and Biopharm, 15, 657-680.

Steinijans VW, Diletti, E. Statistical Analysis of Bioavailability Studies: Parametric and Nonparametric Confidence Intervals. Eur J Clin Pharmacol, 1983;24:127-136.

# 14. ATTACHMENTS

# 14.1. Table of Contents for Data Display Specifications

For the Clinical Pharmacology Study Report the following section numbering will apply:

Section 8: Study Population

Section 9: Safety

Section 10: Pharmacokinetic

Section 11: Pharmacodynamic / Biomarker

Section 12: Pharmacogenetics Analysis

Listed below are the planned figures, tables and listings to be produced for inclusion in the 200942 clinical study report:

IDSL standard displays beginning with "CP\_" are specific to Clinical Pharmacology and can be found in the IDSL database under "Supporting Documentation -> TST use of IDSL Core Choices -> ClinPharm -> All -> Clin Pharm Options for Statistical Displays".

# 14.1.1. Study Population

| Table No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 9.1 | All Subjects | ES1a | Summary of Subject Disposition | By Cohorts and both combined | QSI (Prog) | SAC |
| 9.2 | All Subjects | DM1 | Summary of Demographic<br>Characteristics | By Cohorts and both combined 2.Add BMI, Weight Height, | QSI (Prog) | SAC |
| 9.3 | All Subjects | DM5 | Summary of Race and Racial Combinations | By Cohorts and both combined | QSI (Prog) | SAC |
| 9.4 | All Subjects | DM6 | Summary of Race and Racial Combinations Details | By Cohorts and both combined | QSI (Prog) | SAC |
| 9.5 | Enrolled | NS1 | Summary of Number of Subjects by Country and Site ID | By Cohorts and both combined | QSI (Prog) | SAC |
| 9.6 | Enrolled | DM11 | Summary of Age Ranges | By Cohorts and both combined | QSI (Prog) | SAC |

# 14.1.2. Safety Tables

# **Tables**

| Table<br>No. | Population | Example Shell | | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.1 | All Subjects | CP_AE1p | Summary of All Adverse Events | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.2 | All Subjects | CP_AE1p | Summary of Drug-Related Adverse Events By Cohorts and both combined QSI (Programmer) | | QSI (Prog) | SAC |
| 10.3 | All Subjects | CP_AE1p | Summary of Serious Adverse Events | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.4 | All Subjects | CP_AE1p | Summary of AEs Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.5 | All Subjects | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.6 | All Subjects | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.7 | All Subjects | LB1 | Summary of Haematology Laboratory Values | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.8 | All Subjects | LB1 | Summary of Change from Baseline in Haematology Laboratory Values By Cohorts and both combined | | SAC | |
| 10.9 | All Subjects | LB1 | Summary of Chemistry Laboratory Values | By Cohorts and both combined | QSI (Prog) | SAC |

| Table<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.10 | All Subjects | LB1 | Summary of Change from Baseline in Chemistry Laboratory Values | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.11 | All Subjects | EG1 | Summary of ECG Findings | By Cohorts and both combined description | QSI (Prog) | SAC |
| 10.11 | All Subjects | EG2 | Summary of ECG Values | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.12 | All Subjects | EG2 | Summary of Change from Baseline in ECG Values | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.13 | All Subjects | VS1 | Summary of Vital Signs | By Cohorts and both combined | QSI (Prog) | SAC |
| 10.14 | All Subjects | VS1 | Summary of Change from Baseline for Vital Signs | By Cohorts and both combined | QSI (Prog) | SAC |

# 14.1.3. Pharmacokinetic Figures and Tables

# **Figures**

| Figure<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.1 | PK | PKCF1p | Individual Plasma GSK1278863 Concentration-Time Plots – by Subjects | x-axis should display Actual relative time Include line for LLQ along with footnote defining LLQ value. Include values below LLQ. | QSI (Prog) | SAC |
| 11.2 | PK | PKCF1p | Individual Plasma GSK2391220 (M2) Concentration-<br>Time Plots – by Subjects | | QSI(Prog) | SAC |
| 11.3 | PK | PKCF1p | Individual Plasma GSK2506104 (M3) Concentration-<br>Time Plots – by Subjects | | QSI(Prog) | SAC |
| 11.4 | PK | PKCF1p | Individual Plasma GSK2487818 (M4) Concentration-<br>Time Plots – by Subjects | | QSI(Prog) | SAC |
| 11.5 | PK | PKCF1p | Individual Plasma GSK2506102 (M5) Concentration-<br>Time Plots – by Subjects | | QSI(Prog) | SAC |
| 11.6 | PK | PKCF1p | Individual Plasma GSK2531398 (M6) Concentration-<br>Time Plots – by Subjects | | QSI(Prog) | SAC |
| 11.7 | PK | PKCF1p | Individual Plasma GSK2531401 (M13) Concentration-Time Plots – by Subjects | | QSI(Prog) | SAC |

| Figure<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.8 | PK | PKCF4 | Mean (± SD) Plasma GSK1278863 Concentration-Time Plots (Linear and Semi-log) by Cohort | X-axis displays planned relative time Include line for LLQ along with footnote defining LLQ value. Can do both the cohorts in one page by adding legends | QSI (Prog) | SAC |
| 11.9 | PK | PKCF4 | Mean (± SD) Plasma GSK2391220 (M2) Concentration-<br>Time Plots (Linear and Semi-log) by Cohort | Can do both the cohorts in one page by adding legends | QSI(Prog) | SAC |
| 11.10 | PK | PKCF4 | Mean (±SD) Plasma GSK2506104 (M3) Concentration-<br>Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.11 | PK | PKCF4 | Mean (±SD) Plasma GSK2487818 (M4) Concentration-<br>Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.12 | PK | PKCF4 | Mean (±SD) Plasma GSK2506102 (M5) Concentration-<br>Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.13 | PK | PKCF4 | Mean (±SD) Plasma GSK2531398 (M6) Concentration-<br>Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.14 | PK | PKCF4 | Mean (±SD) Plasma GSK2531401 (M13)<br>Concentration-Time Plots (Linear and Semi-log) by Cohor | t | QSI(Prog) | SAC |

| Figure<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.15 | PK | PKCF5 | Median (range) Plasma GSK1278863 Concentration-Time Plots (Linear and Semi-log) by Cohort | 1. Include bars for range. 2. X-axis displays planned relative time. 3. Include line for LLQ along with footnote defining LLQ value. 3. Can do both the cohorts in one page by adding legends | QSI (Prog) | SAC |
| 11.16 | PK | PKCF5 | Median (range) Plasma GSK2391220 (M2) Concentration-Time Plots (Linear and Semi-log) by Cohort | Can do both the cohorts in one page by adding legends | QSI(Prog) | SAC |
| 11.17 | PK | PKCF5 | Median (range) Plasma GSK2506104 (M3) Concentration-Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.18 | PK | PKCF5 | Median (range) Plasma GSK2487818 (M4) Concentration-Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.19 | PK | PKCF5 | Median (range) Plasma GSK2506102 (M5) Concentration-Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.20 | PK | PKCF5 | Median (range) Plasma GSK2531398 (M6) Concentration-Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 11.21 | PK | PKCF5 | Median (range) Plasma GSK2531401 (M13) Concentration-Time Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |

| Figure<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.22 | PK | PKCF1p | Individual Plasma GSK1278863 Concentration-Time Plots – by Cohort | Can do both the cohorts in one page by adding legends | QSI(Prog) | SAC |
| 11.23 | PK | PKCF6 | Individual Plasma GSK2391220 (M2) Concentration-<br>Time Plots by Cohort (Linear and Semi-Log) | Can do both the cohorts in one page by adding legends | QSI(Prog) | SAC |
| 11.24 | PK | PKCF6 | Individual Plasma GSK2506104 (M3) Concentration-<br>Time Plots by Cohort (Linear and Semi-Log) | | QSI(Prog) | SAC |
| 11.25 | PK | PKCF6 | Individual Plasma GSK2487818 (M4) Concentration-<br>Time Plots by Cohort (Linear and Semi-Log) | | QSI(Prog) | SAC |
| 11.26 | PK | PKCF6 | Individual Plasma GSK2506102 (M5) Concentration-<br>Time Plots by Cohort (Linear and Semi-Log) | | QSI(Prog) | SAC |
| 11.27 | PK | PKCF6 | Individual Plasma GSK2531398 (M6) Concentration-<br>Time Plots by Cohort (Linear and Semi-Log) | | QSI(Prog) | SAC |
| 11.28 | PK | PKCF6 | Individual Plasma GSK2531401 (M13) Concentration-Time Plots by Cohort (Linear and Semi-Log) | | QSI(Prog) | SAC |
| 11.29 | PK | PKCF6 | Individual Plasma Concentration-Time Plots by<br>Analyte at Predose (Linear and Semi Log) | | QSI (Prog) | SAC |
| 11.30 | PK | PKCF6 | Mean Plasma Concentration-Time Plots by Analyte at Predose (Linear and Semi Log) | | QSI (Prog) | SAC |
| 11.31 | PK | PKCF6 | Median Plasma Concentration-Time Plots by Analyte at Predose (Linear and Semi Log) | | QSI (Prog) | SAC |

# **Tables**

| Table<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.1 | PK | PKCT1 | Summary of Plasma GSK1278863 and its metabolites Concentration-Time Data | By Cohort and combined Refer Table 1 for Cohort description | QSI(Prog) | SAC |
| 11.2 | PK | PKPT4 | Summary of Derived Plasma Pharmacokinetic<br>Parameters of GSK1278863 and its<br>Metabolites | 1.By Cohort and combined Refer Table 1 for Cohort description | QSI(Prog) | SAC |
| 11.3 | PK | Exhibit 1 | Summary of Analysis Results for Steady-State Pharmacokinetic Profile of Trough concentration (Cτ) for each Metabolite | | QSI(Stat) | SAC |
| 11.4 | PK | Exhibit 2 | Summary of Results of Statistical Analysis of<br>Derived Plasma GSK1278863 Parameters to<br>Assess Accumulation for each Metabolite | | QSI(Stat) | SAC |
| 11.5 | PK | Exhibit 3 | Summary of Results of Statistical Analysis of<br>Derived Plasma GSK1278863 Parameters to<br>Assess Time Invariance for each Metabolite | | QSI(Stat) | SAC |
| 11.6 | PK | PKCT1 | Summary of Percent Protein Bound of Plasma GSK1278863 and select metabolites | | QSI (Stat) | SAC |

# 14.1.4. Pharmacodynamic Figures and Tables

# **Figures**

| Figure<br>No. | Population | IDSL No. /<br>Example Shell | Title | Programming Notes | Responsibility | Priority |
|---|---|---|---|---|---|---|
| 12.1 | Subjects Concentration-Time Plots – by Subjects | | x-axis should display Actual relative time Include line for LLQ along with footnote defining LLQ value. Include values below LLQ. | QSI (Prog) | SAC | |
| 12.2 | All<br>Subjects | PKCF1p | ndividual Hepcidin Concentration-Time Plots - by Subjects | | QSI(Prog) | SAC |
| 12.3 | All<br>Subjects | PKCF4 | Mean (±SD) Plasma Erythropoietin Concentration-Time Plots (Linear and Semilog) by Cohort 1. X-axis displays planned relative time 2. Include line for LLQ along with footnote defining LLQ value. | | QSI (Prog) | SAC |
| 12.4 | All<br>Subjects | PKCF4 | Mean (±SD) Hepcidin Concentration-Time<br>Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |
| 12.5 | All<br>Subjects | PKCF5 | Median (range) Plasma Erythropoietin<br>Concentration-Time Plots (Linear and Semilog) by Cohort | Include bars for range. X-axis displays planned relative time. Include line for LLQ along with footnote defining LLQ value. | QSI (Prog) | SAC |
| 12.6 | All<br>Subjects | PKCF5 | Median (range) Hepcidin Concentration-Time<br>Plots (Linear and Semi-log) by Cohort | | QSI(Prog) | SAC |

| Figure<br>No. | Population | IDSL No. /<br>Example Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 12.7 | All<br>Subjects | PKCF6 | Individual Plasma Erythropoietin<br>Concentration-Time Plots by Cohort (Linear<br>and Semi-Log) | | QSI(Prog) | SAC |
| 12.8 | All<br>Subjects | PKCF6 | Individual Hepcidin Concentration-Time Plots by Cohort (Linear and Semi-Log) | | QSI(Prog) | SAC |

# **Tables**

| Table No. | Population | IDSL No. /<br>Example Shell | Title | Additional<br>Programming<br>Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 12.1 | All Subjects | PKPT 4 | Summary Statistics of Hepcidin and Erythropoietin | By Cohort and both combined | QSI (Prog) | SAC |

# 14.1.5. ICH Listings

| Table<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 1 | All Subjects | DM2 | Listing of Demographic Characteristics | By Cohorts 2. Add BMI, Weight ,Height, | QSI(Prog) | SAC |
| 2 | All Subjects | DM9 | Listing of Race | By Cohorts | QSI(Prog) | SAC |
| 3 | All Subjects | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | By Cohorts | QSI(Prog) | SAC |
| 4 | All Subjects | DV2 | Listing of Protocol Deviations | By Cohorts | QSI (Prog) | SAC |
| 5 | All Subjects | ES2 | Listing of Reasons for Withdrawal By Cohorts QS | | QSI(Prog) | SAC |
| 6 | All Subjects | CP_CM3 | Listing of Concomitant Medication by Generic Term | By Cohorts | QSI(Prog) | SAC |
| 7 | All Subjects | EX3 | Listing of Exposure data | By Cohorts | QSI(Prog) | SAC |
| 8 | All Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | By Cohorts | QSI(Prog) | SAC |
| 9 | All Subjects | CP_AE8 | Listing of All Adverse Events | By Cohorts | QSI(Prog) | SAC |
| 10 | All Subjects | CP_AE8a | Listing of SAE | By Cohorts | QSI(Prog) | SAC |
| 11 | All Subjects | CP_AE8 | Listing of AE leading to Withdrawal | Listing of AE leading to Withdrawal By Cohorts QSI(Prog) | | SAC |
| 12 | All Subjects | CP_LB5 | Listing of Haematology Abnormalities of Potential By Cohorts QSI(Prog) Clinical Importance | | SAC | |
| 13 | All Subjects | CP_LB6 | Listing of all Hemeatology Laboratory Data for<br>Subjects with PCI Abnormalities | By Cohorts | QSI(Prog) | SAC |

| Table<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Progra | mming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|---|
| 14 | All Subjects | CP_LB5 | Listing of Chemistry Abnormalities of Potential Clinical Importance | By Coh | orts | QSI(Prog) | SAC |
| 15 | All Subjects | CP_LB6 | Listing of all Clinical Chemistry laboratory Data for subjects with PCI abnormalities By Cohorts | | QSI(Prog) | SAC | |
| 16 | All Subjects | CP_EG5 | Listing of Abnormal ECG findings | ing of Abnormal ECG findings By Cohorts | | QSI(Prog) | SAC |
| 17 | All Subjects | CP_EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | By Cohorts | | QSI(Prog) | SAC |
| 18 | All Subjects | CP_VS4 | Listing of Vital Signs of Potential Clinical Importance | By Cohorts | | QSI(Prog) | SAC |
| 19 | All Subjects | CP_VS4 | Listing of all Vital Signs for subjects with any value of Potential Clinical Importance | By Coh | orts | QSI(Prog) | SAC |
| | onal Displays: The ment forms have | | olays will only be produced when a liver event has occurred. | ed, as def | ined in the study | protocol, and the Liv | er Event |
| 20 | All Subjects | LIVER5 | Listing of Liver Events in Relation to Time of Treatment | t | By Cohorts | QSI(Prog) | SAC |
| 21 | All Subjects | LIVER6 | Listing of Liver Event Information for RUCAM Score | | By Cohorts | QSI (Prog) | SAC |
| 22 | All Subjects | LIVER7 | Listing of Liver Biopsy Details | | By Cohorts | QSI (Prog) | SAC |
| 23 | All Subjects | LIVER8 | Listing of Liver Imaging Details | | By Cohorts | QSI (Prog) | SAC |

# 14.1.6. Other Listings

| Table<br>No. | Population | IDSL No. /<br>Example<br>Shell | Title | Programming Notes | Responsibility | Delivera<br>ble<br>Priority |
|---|---|---|---|---|---|---|
| 1 | All Subjects | AE2 | Relationship between System Organ Class and Verbatim Text | By Cohorts | QSI(Prog) | SAC |
| 2 | PK | PKCI1P | Listing of Plasma GSK1278863 and Metabolite Pharmacokinetic Concentration-Time Data | By Cohorts | QSI(Prog) | SAC |
| 3 | PK | PKPL1P | Listing of Derived Plasma Pharmacokinetic Parameters of GSK1278863 and its Metabolites | By Cohorts | QSI(Prog) | SAC |
| 4 | PK | PHI113635/Li<br>sting 31 | Listing of effluent Peritoneal Dialysis Fluid Data | By Cohorts | QSI(Prog) | SAC |
| 5 | All Subjects | PHI113635/Li<br>sting 31 | Listing of Hepcidin and Erythropoietin | By Cohorts | QSI(Prog) | SAC |
| 6 | PK | | Raw SAS Output for Summary of Analysis Results for Steady-State Pharmacokinetic Profile of Trough concentration (Cτ) | | QSI(Stat) | SAC |
| 7 | PK | | Raw SAS Output for Summary of Results of Statistical Analysis of Derived Plasma GSK1278863 Parameters to Assess Accumulation | | QSI(Stat) | SAC |
| 8 | PK | | Raw SAS Output for Summary of Results of Statistical Analysis of Derived Plasma GSK1278863 Parameters to Assess Time Invariance | | QSI(Stat) | SAC |
| 9 | PK | | Raw SAS Output for Summary Analysis Results for Comparison of Pharmacokinetic Parameters of GSK1278863 and its Metabolites using ANOVA | | QSI(Stat) | SAC |

200942

# 14.2. Data Display Specifications (Example Shells)

Example : Exhibit 1 Page 1 of n

Protocol: 200942

Population : PK Population

Table xx.x Summary of Results of Statistical Analysis to Assess Steady state

| Da | y Back-7 | Transformed Slope | 90% Confidence Interval |
|----|----------|-------------------|-------------------------|
| 1- | -14 1 | . 0.5 | 1.03, 1.08) |

200942

Example : Exhibit 2 Page 1 of n
Protocol : 200942

Population : PK Population

Table x.x Summary of Results of Statistical Analysis to Estimate Accumulation Ratio

| Parameter | Comparison | Geom.LsMean | | | Ratio | 90%<br>Confidence Interval |
|---|---|---|---|---|---|---|
| | - | | | | | |
| | | n | Test | n Ref | | |
| AUC(0-t)(pg*hr/mL) | Day 14 vs Day 1 | 12 | 0.910 | 12 0.780 | 1.166 | ( 0.843, 0.978 ) |

200942

Example : *Exhibit3*Protocol : 200942

Page 1 of n

Population : PK Population

Table x.x Summary of Results of Statistical Analysis to Estimate Time Invariance

| Comparison | | Geom.Ls | Mean | Ratio | 90% |
|---|---|---|---|---|---|
| | | | | | Confidence Interval |
| | n | Test | n Ref | | |
| AUC(0-τ)Day 14 vs AUC(0-∞)Day 1 | <br>12 | 0.910 | 12 0.780 | 1.166 | ( 0.843, 0.978 ) |